CLINICAL TRIAL: NCT01980381
Title: Treatment of Depression and/or Anxiety - a Randomized Clinical Trial of the Tree Theme Method® (TTM) as an Intervention
Brief Title: Treatment of Depression and/or Anxiety - the Tree Theme Method® (TTM) as an Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kronoberg County Council (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LTK/120995
Record Dates: First submitted 2013-08-06; First posted 2013-11-11 (Estimated); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Depression; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tree Theme Method ® (TTM) intervention (Experimental): The TTM involves storytelling and story making, in which the patient draws tree maps representing certain periods of his/her life.
  Interventions: Other: Tree Theme Method ® (TTM)
- Control group (No Intervention): Treatment as usual, with focus on the present everyday occupations

INTERVENTIONS:
Other: Tree Theme Method ® (TTM) — The TTM method is based on creative activities and occupational life story telling, implies that the paints trees representing different life periods, looking back and forward, as well as the present.
  Arms: Tree Theme Method ® (TTM) intervention

SUMMARY:
Depression and anxiety are among our most common diseases and the prevalence is increasing. When suffering from depression or anxiety, the individual's ability to cope with everyday life occupations is decreased, as well as the ability to relate to others. The Tree Theme Method® (TTM) is a treatment method. The purpose is to enhance the ability to develop strategies for occupations in everyday life and relationships with others. The method involves using creative activities to create a life story focusing on everyday occupations and to create an imagination of future possibilities/goals. The TTM is a short-term therapy with five sessions. The treatment also implies that the patient is asked to identify various homework tasks to perform between the sessions.

The aim of the project is to investigate the effects of the TTM compared to a control group for people with depression and anxiety diagnosis. The intention is to examine the effect on outcome measures regarding psychological symptoms, everyday occupations and health. The study has been approved by the Regional Ethical Review Board.

The project is a randomized multicenter study with an intervention group and a control group. A total of 130 patients will be included. Inclusion criteria are patients with depression and/or anxiety in the age of 18-65 years and who have problems with their everyday occupations. Exclusion criteria are individuals with a severe somatic illness or psychosis and/or who have difficulties to understand and fill out self-rating questionnaires.

The project implies that doctors will refer appropriate patients to the occupational therapist. After informed consent each patient will be drawn to the TTM or control. Before and after the treatment, as well as 3 and 12 months after finished treatment the patient will meet a project assistant in order to respond to questionnaires regarding psychological symptoms, everyday occupations and health.

The study is a collaborative project involving the Region Skåne, Kronoberg County Council, and Jönköping County Council. Doctors will recruit patients and occupational therapists will perform the treatment. The research team comprise of researchers from Kronoberg County Council (B Gunnarsson and K Hedin), Lund University (C Håkansson) and School of Health Sciences in Jönköping (P Wagman).

ELIGIBILITY:
Inclusion Criteria:

* Depression and/or anxiety in age of 18-65 years and problems with everyday occupations.

Exclusion Criteria:

* Severe somatic illness or psychosis and/or difficulties to understand and fill out self-rating questionnaires

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2013-01; Primary Completion 2025-01 (Actual); Study Completion 2025-07 (Actual)

PRIMARY OUTCOMES:
Psychological symptoms | Change from baseline to after treatment (6-9 weeks), 3 and 12 months
  Psychological symptoms measured by the SCL-90-R(Derogatis, 1992) Depression measured by the MADRS-S(Montgomery & Åsberg, 1979) Anxiety/depression measured by the HAD(Zigmond & Snaith, 1983)

SECONDARY OUTCOMES:
Everyday occupations | Change from baseline, after treatment (6-9 weeks), and 3 and 12 months
  Everyday occupations measured by the Occupational performance and satisfaction with occupational performance measured (COPM)(Law et al., 1998), the Satisfaction with Daily occupations (SDO)(Eklund, 2004)and the Occupational balance (Wagman, Håkansson & Björklund, 2011).

CONTACTS AND LOCATIONS:
Overall Officials: Birgitta A Gunnarsson, PhD, Study Chair — Kronoberg CC
Locations (1):
- Kronoberg County Council, Vaxjo, Kronoberg County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Eklund M, Gunnarsson AB. The relevance of employing a three-perspective view on occupational balance among people with depression and/or anxiety disorders. Scand J Occup Ther. 2025 Mar 6;32(1):2474853. doi: 10.1080/11038128.2025.2474853. Epub 2025 Mar 19. PMID 40104977
- [Derived] Birgitta Gunnarsson A, Wagman P, Hedin K, Hakansson C. Treatment of depression and/or anxiety - outcomes of a randomised controlled trial of the tree theme method(R) versus regular occupational therapy. BMC Psychol. 2018 May 23;6(1):25. doi: 10.1186/s40359-018-0237-0. PMID 29792226
- [Derived] Gunnarsson AB, Wagman P, Hakansson C, Hedin K. The Tree Theme Method(R) (TTM), an occupational therapy intervention for treating depression and anxiety: study protocol of a randomized controlled trial. BMC Psychol. 2015 Nov 9;3:40. doi: 10.1186/s40359-015-0097-9. PMID 26552426